CLINICAL TRIAL: NCT03999697
Title: Clinical Study of CD22 CAR T Cells in the Treatment of Patients With Relapsed or Refractory CD22 Positive B Cells With Acute Lymphoblastic Leukemia
Brief Title: A Clinical Research of CD22-Targeted CAR-T in B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-22-I-001
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Primary Cutaneous Follicle Centre Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Mantle Cell Lymphoma; Plasma Cell Neoplasm; B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Neoplasms, Plasma Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-CD22 Cell immunotherapy (Experimental): Enrolled patients will receive CAR-CD22 cell immunotherapy with a novel specific chimeric antigen receptor targeting CD22 antigen by infusion.
  Interventions: Drug: Autologous chimeric antigen receptor T cell transfusing agent targeting CD22

INTERVENTIONS:
Drug: Autologous chimeric antigen receptor T cell transfusing agent targeting CD22 — The enrolled patients will receive autologous-derived CD22-targeted CAR-T cells in 1 day with 100% of the total expected dosage after receiving lymphodepleting chemotherapy

SUMMARY:
Evaluation of the efficacy and safety of CD22-targeted chimeric antigen receptor T(CAR-T) cells in the treatment of recurrent or refractory CD22 positive B cell acute lymphoblastic leukemia (B-ALL)

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with CD22+ B cell malignancies in patients who have no available curative treatment options except stem cell transplantation, with limited prognosis (several months to < 2 year survival) and no available treatment option to achieve complete remission prior to transplant. Some patients who have enrolled to other CD22-CAR-T cell therapy trials may be eligible if their CD22-CAR-T cells cannot be produced successfully because they have insufficient T cells to allow the CD22-CAR-T cells to be made; their T cells are inefficiently transduced with CAR viruses; or their CAR-T cell expansion is failed. All of those patients must meet the following criteria:

1. Eligible diseases: Acute lymphocytic leukemia (ALL), Chronic lymphocytic leukemia (CLL), Follicular lymphoma, Mantle cell lymphoma, B-cell prolymphocytic leukemia, and diffuse large cell lymphoma, previously identified as CD22+.
2. Patients 3 years of age or older, and must have a life expectancy > 12 weeks.
3. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
4. Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR CD22 cells.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
6. Ability to give informed consent.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) involvement.
2. Pregnant or nursing women may not participate.
3. Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. Previously treatment with any gene therapy products.
7. The existence of unstable or active ulcers or gastrointestinal bleeding.
8. Patients with a history of organ transplantation or are waiting for organ transplantation.
9. Patients need anticoagulant therapy (such as warfarin or heparin).
10. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events That Are Related to Treatment | 2 years
  Determine the toxicity profile of the CD22 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.03
The effect after treatment | 24 weeks
  ORR within 24 weeks after infusion （CR+CRi）

SECONDARY OUTCOMES:
In vivo existence of Anti-CD22 CAR-T cells | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen·Anke cellular therapeutics Co., Ltd, Hefei, Anhui, China